CLINICAL TRIAL: NCT05210010
Title: A Prospective Study to Assess the Utility of CA-4F in a Canadian Cardiology Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ensho Health Intelligent Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SA001401001
Record Dates: First submitted 2021-12-30; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Transthyretin Amyloid Cardiomyopathy ("ATTR-CM")

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Algorithm (Other): All participating cardiologists.
  Interventions: Device: CA-4F

INTERVENTIONS:
Device: CA-4F — The study intervention is the CA-4F algorithm developed by Ensho Health.
  The algorithm is a process for converting input parameters to a CA-4F Risk Score intended to facilitate clinical prioritization of patients suitable for follow-up investigation for ATTR-CM.
  The algorithm is applied using the CA-4F Likelihood Estimator which encodes it in software and records its outputs. The CA-4F Likelihood Estimator is controlled through a graphical user interface called the CA-4F Controller.
  The CA-4F Likelihood Estimator and its Controller are Class I medical devices in Canada registered under the Medical Device Establishment License of Ensho Health (license 16208).

SUMMARY:
This study will assess whether CA-4F can improve diagnosis of ATTR-CM in a community cardiology setting when used to screen electronic medical record data for patients suitable for follow-up investigations.

DETAILED DESCRIPTION:
This is a prospective multicentre observational study to assess whether CA-4F can improve diagnosis of ATTR-CM in a community cardiology setting when used to screen electronic medical record data for patients suitable for follow-up investigations.

The algorithm will be used to screen electronic health records of participating cardiologists for patients suitable for PYP scans to investigate potential ATTR-CM and determine its positive predictive value.

Input parameters to the algorithm will be extracted from the pseudonymized electronic health records of patients who visited participating cardiologists in the 12 months preceding their enrolment.

The records of patients with elevated pre-test likelihood of ATTR-CM will be queried for Canadian Heart Failure Society red flag symptoms to facilitate clinical review. Participating cardiologists will review the red flag symptoms and electronic health records of patients with elevated pre-test likelihoods and document whether further investigation with PYP is clinically justified with supporting rationale.

Patients for which further investigation is clinically justified will be referred for confirmatory testing and the results of additional investigations will be documented. The positive predictive values of "moderate", "high" and "very high" CA-4F Risk Scores will be calculated by determining the percentage of those patients for which further investigations were performed and resulted in diagnosis of ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

* Licensed cardiologist in the Canadian provinces of Ontario, Saskatchewan or British Columbia
* Outpatient cardiology practice with ≥1,200 unique patients annually
* Have used an electronic medical record system for ≥36 months from enrollment
* Currently subscribed to the Advanced Computing Platform by Ensho Health or using a cloud-hosted electronic medical record system compatible with the Apollo Electronic Data Capture System
* Experience with the clinical management of ATTR-CM
* Access to PYP scanning for follow-up investigations
* Previous participation in clinical studies

Exclusion Criteria:

* Predominantly hospital-based cardiology practice
* Have used an electronic medical record system for <36 months from enrollment
* Electronic medical record system incompatible with the Apollo Electronic Data Capture system
* No prior experience with the clinical management of ATTR-CM
* No access to PYP scanning for follow-on investigations
* No prior participation in clinical studies

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical utility of CA-4F | Six months
  Positive predictive value of "moderate" or greater CA-4F Risk Score as confirmed by PYP scan

SECONDARY OUTCOMES:
Optimal threshold for clinical use | Six months
  Positive predictive values of "moderate," "high," "very high," and "high" or greater CA-4F Risk Scores as confirmed by PYP scan

OTHER OUTCOMES:
Impacts of CA-4F on age at first diagnosis | Six months
  Difference in age at diagnosis of patients diagnosed through the study and patients of participating cardiologists previously diagnosed with ATTR-CM
Impacts of CA-4F on rate of diagnosis in priority subgroups | Six months
  Difference in biological sex distribution and left ventricular wall thickness measurements of patients diagnosed through the study and patients of participating cardiologists previously diagnosed with ATTR-CM

CONTACTS AND LOCATIONS:
Overall Officials: Taha Bandukwala, MD, Principal Investigator — Chief Medical Officer
Locations (3):
- Canada (3):
  - Site 85237, North Vancouver, British Columbia
  - Site 26174, Oakville, Ontario
  - Site 47844, Scarborough Village, Ontario